CLINICAL TRIAL: NCT02020746
Title: A Multicenter, International, Prospective, Randomized, Vehicle Controlled, Assessor Blinded Study Performed in Subjects With Hard to Heal Wounds, to Evaluate the Efficacy and Safety of Enzymatic Debridement With EscharEx
Brief Title: Efficacy and Safety Study of EscharEx to Treat (Debride) Hard to Heal Wounds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MW 2013-07-10
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hard to Heal Wounds; Venous Leg Ulcers; Diabetic Lower Extremity Ulcers; Traumatic/ Post Operative Wounds
MeSH Terms: interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- EscharEx (Active Comparator): Enzymatic debridement
  Interventions: Drug: EscharEx
- Gel Vehicle (Placebo Comparator): Control arm
  Interventions: Drug: Gel Vehicle

INTERVENTIONS:
Drug: EscharEx
  Arms: EscharEx
Drug: Gel Vehicle
  Arms: Gel Vehicle

SUMMARY:
The main objective of this study is to assess the safety and the efficacy of EscharEx in preparing the wound's bed in patients with hard to heal venous leg ulcers, diabetic lower extremity ulcers and traumatic/post operative wounds.

This study will be a multi-center, assessor blinded, randomized, controlled study intended to demonstrate superiority of EscharEx debriding treatment over the Gel Vehicle control treatment in patients with hard to heal wounds.

72 + 24 adults with >50% necrotic/slough/fibrin non-viable tissue on a hard to heal wound (venous leg ulcer, diabetic lower extremity ulcer or traumatic/ post operative wound) between 5 cm2 and 200 cm2 (surface area in stage 1) or 3 cm2 - 150 cm2 (in stage 2), will be enrolled into the study.

Patients will undergo a 1 week screening period (2 visits) which will include: record of demographics, medical history and concomitant medications, vital signs, physical examination, clinical laboratory tests, wound photography and assessments and questionnaires (wound status and quality of life). During this period wounds will be treated by standard treatment per the decision of the physician. During this screening period, subjects whose study wound size (surface area) decreases by more than 20 percent will be excluded. Following completion of the screening process, eligible patients will be randomized to either EscharEx or Gel vehicle debridement treatments. In stage 1 (72 patients): Treatment will be performed for up to 10 applications or until complete debridement is achieved, whichever occurs first. In stage 2 (24 patients): Treatment will be performed for up to 8 applications or until complete debridement is achieved, whichever occurs first. Following each application the wound will be washed, photographed and assessed for wound size, removal of nonviable tissue and change in granulation tissue (by digital planimetry software), wound status, and safety parameters. Subsequent to each debridement treatment the wound will be dressed with moist-to-moist saline gauze (except when successive 24h or 48h treatments are performed, in the second stage). Following completion of the debridement treatment period, patients will be treated according to standard procedures and evaluated (wound assessments) once a week until complete wound closure for up to 12 weeks from last application (up to 12 visits). Only during the first stage of the study, for patients who achieved wound closure, additional 3 monthly (3 visits) follow- up visits of wound closure recurrence will be conducted. Quality of life (QoL) will be evaluated at the last follow-up visit - 3 months post wound closure follow-up period. For patients who didn't achieve wound closure only the 3 months FU visit will be conducted. For patients enrolled at the second stage, if wound closure was achieved at the 12 weeks follow-up, additional visit will be performed 2 weeks later to confirm wound closure.

ELIGIBILITY:
Inclusion Criteria

* Patients, men or women, are between 18 and 90 years of age.
* Patient with venous leg ulcer or diabetic (lower extremity) ulcer or traumatic/post operative wound (determined by medical history and physical examination)
* Wound is not healing for at least 4 weeks
* The necrotic/slough/fibrin non-viable tissue area is at least 50% of wound area (assessed by clinical evaluation)
* Wound surface area is in the range of 5- 200 cm2 in the first stage and 3 - 150cm2 in the second stage.
* Patient understands the nature of the procedure, able to adhere to the protocol regimen, and provides written informed consent prior to any study procedure
* The Wound is classified as a wound involving full skin thickness but not penetrating to cavities or open joint spaces

Exclusion Criteria

* Evidence of active osteomyelitis of target organ,
* Patients with more than one hard to heal wounds wounds which require debridement and with an area greater than or equal to 2cm2,
* Presence of purulent discharge, deep-tissue abscess, cellulitis or tissue damage extending >2 cm around the wound's edge, gangrene or signs of systemic infection,
* Wound size decreased by > 20% after 1 week of standard-of-care-only period (screening period),
* Patients with pre-enrolment wounds which are covered by eschar heavily saturated with iodine or by Silver sulfadiazine (SSD) pseudoeschar (e.g. pseudoeschar as a result of SSD treatment),
* Ankle-Brachial Index (ABI) ≤ 0.7 or a significant decrease in the blood flow of the extremity as demonstrated by US doppler.
* Wound has sinus tracts or tunnels extending under healthy tissue,
* Patients undergoing renal or peritoneal dialysis,
* Recent history (less than 4 weeks) of myocardial infarction (MI) or concurrent acute injury or disease that might compromise the patient's welfare,
* Any condition that would preclude safe participation in the study: evidence of significant hematological (severe pre-existing coagulation disorder), cardiovascular, liver or neoplastic disease, or any other immediate life threatening condition,
* Patient is currently receiving, or has received at any time within one month prior to enrollment, any medications or treatments known to affect the wound healing processes; these include: chronic systemic steroid intake with topical skin changes (thin, fragile with multiple hematomas and previous laceration history, immuno-suppressive drugs, radiation therapy and chemotherapy.
* History of allergy or atopic disease or a known sensitivity to pineapples, papaya, bromelain or papain,
* Pregnant women (positive pregnancy test) or nursing mothers,
* Participation in another investigational drug trial within 30 days prior to enrollment or anticipated participation while enrolled in the study,
* Concurrent use of non-approved drugs or alcohol abuse.
* Patients with poor nutritional status (albumin < 2.5g/dl), poor diabetic control (HbA1c > 12%), anemia (hemoglobin<8 g/dL), a leukocyte counts < 4,000// μl or >15000/μl, abnormal liver function (AST, ALT>2 x upper limit of normal range), renal failure (Cr > 3 mg/dl);
* Mentally incapacitated adults who are incapable of giving legal consent (e.g. dementia, psychiatric patients, etc),
* Patients with general skin disorders (Psoriasis, Panniculitis, ect) that might deteriorate as a result of local trauma.
* Patients with skin disorders unrelated to the wound that are presented adjacent to the wound
* Clinical suspicion of skin cancer associated with the wound (e.g, BCC, SCC), which was not ruled out by biopsy Patients with diagnosed Sepsis during screening phase,
* Patients suffering from Idiopathic Pruritus.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Incidence of complete debridement (non-viable tissue removal) at the end of the debridement period assessed by the blinded assessor by clinical evaluation. | up to 10 treatment days

SECONDARY OUTCOMES:
Rate of complete wound closure | 12 weeks post debridement

CONTACTS AND LOCATIONS:
Locations (8):
- Israel (8):
  - Emek, Afula
  - Rambam MC - Plastic surgery ward, Haifa
  - Meir MC, Kfar Saba
  - Galilee, Nahariya
  - HaSharon hospital, Rabin MC, Petah Tikva
  - Sheba MC, Ramat Gan
  - Kaplan, Rehovot
  - Assaf HaRofeh, Zrifin